CLINICAL TRIAL: NCT01051206
Title: The Effect of 6% Hydroxyethyl Starch 130/0.4 on Blood Loss and Coagulation in Patients Medicated With Antiplatelet Agents Prior to Off-Pump Coronary Bypass Graft Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Jae Kwang Shim, Assistant Professor of Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea
Purpose: Prevention
Other Study IDs: 4-2009-0057
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Occlusive Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 6% hydroxyethyl Stach 130/0.4 — After dividing patients medicated with HES 130/0.4(maximum 33ml/kg/day) during surgery and one day after from the surgery with patients medicated with crystalloid only, compare the effect on the volume of bleeding, blood transfusion, and blood coagulation when using IV fluid.

SUMMARY:
HES 130/0.4 significantly solution will not affect on coagulation and blood loss in patients medicated with antiplatelet agents prior to off-pump coronary bypass surgery (OPCAB).

ELIGIBILITY:
Inclusion Criteria:

* Eighty patients undergoing OPCAB, who were exposed to anti platelet agents until 5 days prior to surgery were randomly allocated to infuse HES 130/0.4 up to 30 ml/kg and followed crystalloid infusion or infuse crystalloid only during perioperative period,

Exclusion Criteria:

Patient who has

* Valvular disease of heart
* MI within 3 months,patient under 40% of left ventricle preoperative output
* left main artery stenosis
* anemia (hemoglobin < 12 g/dl), coagulopathy (Platelet < 100/nl, activated partial thromboplastin time, aPTT) > 80sec, serum creatinine > 1.2 mg/dl, respiratory disease(asthma, COPD, PaO2 < 70 mmHg, pulmonary hypertension or pulmonary edema, etc)
* not consented to this trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
TEG, hemoglobin, platelet count, prothrombin time (PT), partial prothrombin time (aPTT), blood loss, amount of transfusion, urine output, comparing the record data of IV fluid consumption | Preoperative thromboelastography (TEG) and other coagulation variables were measured and follow up data were collected at immediate postoperatively and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea